CLINICAL TRIAL: NCT02698345
Title: Korean Multicenter Prospective Registry of In.PACT DEB for Isolated Popliteal Artery Disease (K-POP Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2015-0081
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Popliteal Artery Disease
Keywords: Popliteal artery disease, drug-eluting balloon, angioplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- K-POP: Patients with isolated popliteal artery disease undergoing endovascular therapy using drug-eluting balloon (In.PACT Admiral, Medtronic)
  Interventions: Device: drug-eluting balloon (In.PACT Admiral, Medtronic)

INTERVENTIONS:
Device: drug-eluting balloon (In.PACT Admiral, Medtronic)

SUMMARY:
* Prospective, multi-center, single-arm registry study
* A total of 100 subjects with isolated popliteal artery lesions according to inclusion and exclusion criteria will be enrolled.
* All popliteal artery lesions will be treated with drug-eluting balloon (In.PACT Admiral, Medtronic). • Atherectomy or use of bare nitinol stent in combination with drug-eluting balloon is allowed • Patients will be followed clinically for 12 months after the procedure.
* Imaging study (Duplex ultrasound, CT angiography or catheter angiography) follow-up will be performed at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years or older
2. Symptomatic peripheral artery disease:

   * Moderate or severe claudication (Rutherford category 2 or 3)
   * Critical limb ischemia (Rutherford category 4 or 5)
3. Atherosclerotic popliteal artery disease (stenosis > 50%)
4. Patients with signed informed consent

Exclusion Criteria:

1. Acute critical limb ischemia
2. Severe critical limb ischemia (Rutherford category 6)
3. Involvement of SFA disease with stenosis
4. Continous total occlusion of all proximal infrapopliteal arteries (origin of the anterior tibial artery or tibioperoneal trunk).
5. Known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, or contrast agent
6. Age > 85 years
7. Severe hepatic dysfunction (> 3 times normal reference values)
8. Significant leucopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
9. LVEF < 40% or clinically overt congestive heart failure
10. Pregnant women or women with potential childbearing
11. Life expectancy <1 year due to comorbidity
12. Previous bypass surgery or stenting for the target popliteal artery
13. Untreated inflow disease of the ipsilateral pelvic or femoropopliteal arteries (more than 50% stenosis or occlusion)

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with isolated popliteal artery disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate | 12 months after the index procedure
  absence of restenosis >50% based on an imaging study (Duplex ultrasound, CT angiography or catheter angiography) at 12 months

SECONDARY OUTCOMES:
Target vessel revascularization rate | 12 months
  frequency of repeat intervention or surgical treatment due to loss of patency at the target vessel

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park JI, Ko YG, Lee SJ, Ahn CM, Rha SW, Yu CW, Park JK, Park SH, Lee JH, Kim SH, Lee YJ, Hong SJ, Kim JS, Kim BK, Hong MK, Choi D. Clinical Outcomes After Drug-Coated Balloon Treatment in Popliteal Artery Disease: K-POP Registry 12-Month Results. Korean Circ J. 2024 Aug;54(8):454-465. doi: 10.4070/kcj.2024.0006. Epub 2024 Apr 29. PMID 38767445